CLINICAL TRIAL: NCT05588999
Title: Comparative Study Between Treatment With Cryotherapy Alone Versus Cryotherapy Plus Salicylic Acid Dressing for Planter Warts
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Dr Mahboob Ali, principal investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHAtd-ETH-38-Derm-22
Record Dates: First submitted 2022-10-11; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Plantar Wart
Keywords: Planter Warts; Cryotherapy; Salicylic Acid
MeSH Terms: interventions — Cryotherapy; Salicylic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Cryotherapy Alone) (Active Comparator): Patients in this Group were subjected to Cryotherapy Alone with liquid nitrogen and received maximum of four treatments given two to three weeks apart
  Interventions: Procedure: Cryotherapy Alone
- Group B (Cryotherapy plus Salicylic Acid) (Active Comparator): Patients in this Group were subjected to cryotherapy plus salicylic acid for a maximum of eight weeks
  Interventions: Combination Product: Cryotherapy plus Salicylic Acid

INTERVENTIONS:
Procedure: Cryotherapy Alone — Patients in Group A were subjected to Cryotherapy Alone with liquid nitrogen and received maximum of four treatments given two to three weeks apart .
  The liquid nitrogen was applied with a spray or a probe
  Arms: Group A (Cryotherapy Alone)
Combination Product: Cryotherapy plus Salicylic Acid — Patients in Group B were subjected to cryotherapy plus with 50% salicylic acid to be properly applied for a maximum of eight weeks The liquid nitrogen was applied with a spray or a probe
  Arms: Group B (Cryotherapy plus Salicylic Acid)

SUMMARY:
Verrucae plantaris (plantar warts) are a frequent cutaneous lesion of the plantar portion of the foot caused by the human papillomavirus (HPV) (HPV).Although HPV is ubiquitous in our environment, cellular and humoral immune responses typically prevent it from spreading or eliminate it.

Warts can be painful and can lead to other difficulties, but there are some populations that are at a higher risk of getting HPV because they encounter the virus more frequently.

In addition to infecting other people, HPV can also spread to other locations in the area. While reducing exposure to risk factors can help prevent plantar wart infection, HPV's widespread nature makes it difficult for such efforts to be effective.

It has been shown in research that plantar warts can spread from person to person through just physical contact with the sores. Warts are more common in people with HPV because the virus disrupts the epithelial barrier. There are over a hundred different forms of the HPV virus, so even though some warts go away on their own after a few years, others may need medical attention.

Warts, according to a number of studies, are extremely common (affecting around 10% of the population) all over the world. More cases of HPV infection have been observed among people under the age of 30, compared to those beyond the age of 30. The estimated prevalence in the United States is between 10% and 20%. However, people with compromised immune systems and those who work with meat are disproportionately at risk.

The cancerous transformation of warts is quite rare. Even while verrucous carcinoma, a malignant form of wart development, is possible, it seldom spreads and only causes localised tissue loss.

Plantar warts are treated in a manner that takes into account the patient's symptoms, personal preferences, and financial situation. Even though there are several therapy options, none of them are particularly effective, and relapses are common after any treatment. As a result, the most accessible and least distressing treatment option should be prioritised.

Since salicylic acid can be used by the patient at home and does not require a doctor's prescription, it is often regarded a first-line therapy for the common wart. It can be as high as 70% effective in curing the disease. Other effective therapies for plantar warts include cryotherapy, retinoic acid, podophyllin, topical 5-fluorouracil, interferon, and imiquimod.

Salicylic acid, in conjunction with cryotherapy, has shown therapeutic efficacy in patients with only foot warts, according to a single prior study. Patients who were given cryotherapy in this trial had a 58% success rate at recovery, whereas those given salicylic acid had a 41% success rate. Hover, there is no discernible statistical difference.

The purpose of this study was to compare the effectiveness of cryotherapy alone against cryotherapy plus salicylic acid dressing for planter warts, keeping in mind the prevalence of treatment for plantar warts and the lack of a well-established, practically applicable, and reliably preventative method in our local population.

ELIGIBILITY:
Inclusion Criteria:

* Patients having aged between 15 to 40 years
* Patients diagnosed with planter warts on toe foot based on clinical and physical examination ,Patients with no history of treatment previously
* Patients of either gender

Exclusion Criteria:

* Patients with impaired healing (such as from diabetes or peripheral vascular disease)
* Immunosuppressed patients
* Patients taking immunosuppressant drugs (such as oral corticosteroids)
* Patients with neuropathy
* Patients receiving renal dialysis
* Patients unable to give informed consent

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
effectiveness of cryotherapy with liquid nitrogen alone and cryotherapy with 50% salicylic acid for the treatment of plantar warts calculated through clinical improvement | 12 weeks
  effectiveness assesed by %clinical improvement=(present % tissue distruction + baseline % tissue destruction)100

CONTACTS AND LOCATIONS:
Locations (1):
- Cmh Abbottabad, Abbottābād, Khyber Pakhtunkhwa, Pakistan